CLINICAL TRIAL: NCT02537899
Title: A Case Series of Patients With Spinal Cord Injury Treated With Standard Therapies and NeuroAiD
Brief Title: Spinal Cord Injury - Assessing Tolerability and Use of Combined Rehabilitation and NeuroAiD
Acronym: SATURN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moleac Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SATURN2015
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Neuroaid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): NeuroAiD
  Interventions: Drug: NeuroAiD

INTERVENTIONS:
Drug: NeuroAiD
  Other Names: MLC601; MLC901

SUMMARY:
SATURN investigates the promising role of NeuroAiD in patients with spinal cord injury and will provide important information on the feasibility of conducting larger controlled trials.

DETAILED DESCRIPTION:
SATURN is a prospective cohort study of patients with moderately-severe to severe spinal cord injury, defined as American Spinal Injury Association Impairment Scale A and B, who are treated with open-label NeuroAiD for 6 months in addition to standard care and followed for 24 months. Anonymized data will be prospectively collected at baseline and months 1, 3, 6, 12, 18, and 24 using a secured online system and will include information on demographics, main diagnostics, neurological and functional state, treatment compliance, concomitant therapies, and side effects, if any.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 to 65 years
* Diagnosed with spinal cord injury between 3 days and 4 weeks
* American Spinal Injury Association Impairment Scale A or B
* Informed consent for inclusion into the database is obtained

Exclusion Criteria:

* Non survivable injury
* Multiple significant trauma (i.e. significant intracranial and extracranial injuries including limb fractures) that would limit observation of recovery from spinal cord injury
* Other conditions that would limit clinical assessment of outcomes (e.g. dementia, demyelinating disease, autoimmune disease, etc)
* Refusal of treatment or contraindication to NeuroAiD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Spinal cord injury severity based on American Spinal Injury Association Impairment Scale | 6 months
Motor recovery based on American Spinal Injury Association Impairment Scale motor score | 6 months
Number of patients experiencing adverse events | 6 months
  Adverse events as individual events and according to organ system, severity, and relatedness

SECONDARY OUTCOMES:
Spinal cord injury severity based on American Spinal Injury Association Impairment Scale | 1, 3, 12, 18, 24 months
Motor recovery based on American Spinal Injury Association Impairment Scale motor score | 1, 3, 12, 18, 24 months
Sensory recovery based on American Spinal Injury Association Impairment Scale sensory score | 1, 3, 6, 12, 18, 24 months
Functional state based on Spinal Cord Independence Measure | 1, 3, 6, 12, 18, 24 months
Quality of life based on Short Form-8 Health Survey | 1, 3, 6, 12, 18, 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Kumar R, Htwe O, Baharudin A, Rhani SA, Ibrahim K, Nanra JS, Gsangaya M, Harun H, Kandar K, Balan M, Peh S, Pokharkar Y, Ingole A, Hisam Ariffin M. Spinal cord injury - assessing tolerability and use of combined rehabilitation and NeuroAiD (SATURN) study - primary results of an exploratory study. J Spinal Cord Med. 2023 Jul;46(4):682-686. doi: 10.1080/10790268.2022.2067972. Epub 2022 May 23. PMID 35604343
- [Derived] Kumar R, Htwe O, Baharudin A, Ariffin MH, Abdul Rhani S, Ibrahim K, Rustam A, Gan R. Spinal Cord Injury-Assessing Tolerability and Use of Combined Rehabilitation and NeuroAiD (SATURN Study): Protocol of An Exploratory Study In Assessing the Safety and Efficacy of NeuroAiD Amongst People Who Sustain Severe Spinal Cord Injury. JMIR Res Protoc. 2016 Dec 5;5(4):e230. doi: 10.2196/resprot.6275. PMID 27919862